CLINICAL TRIAL: NCT06471751
Title: Strengthening Inspiratory and Oropharyngeal Muscles in Moderate Obstructive Sleep Apnea Hypopnea Syndrome
Acronym: REMI SAHOS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Association aide à la recherche médicale de proximité (AIRE) (Unknown); Conseil national de l'ordre des masseurs-kinésithérapeutes (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 23GI019; 2024-A00601-46 (Other: ANSM)
Record Dates: First submitted 2024-06-18; First posted 2024-06-24 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Obstructive Sleep Apnea
Keywords: Inspiratory Muscles Training; Oropharyngeal training
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Inhalation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Strengthening muscles group (Experimental): Home training to strengthen Inspiratory and Oropharyngeal muscles
  Interventions: Other: Inspiratory and Oropharyngeal Muscle Strengthening
- No training group (No Intervention): No intervention

INTERVENTIONS:
Other: Inspiratory and Oropharyngeal Muscle Strengthening — Patients will conduct the training at home, 5 days a week for 3 months. They will perform 2 sets of 30 inspirations against resistance (POWERbreathe® K5 , Powerbreathe International Limited, UK), equal to 70% Maximum Inspiratory Pressure (MIP). Patients will be guided for oropharyngeal exercises.
  The sessions will be supervised by the investigator every 3 weeks. During sessions with the investigator, sessions recorded in the device will be downloaded to verify compliance. A MIP measurement will be performed to adjust the resistance of the device.
  Arms: Strengthening muscles group

SUMMARY:
The Obstructive Sleep Apnea hypopnea Syndrome (OSAS), whose prevalence is 4% of the French population, can lead to serious health consequences (risk of road accidents, onset of cardiovascular disease, etc.). OSAS corresponds to a certain number of interruptions (apneas) or reductions (hypopneas) of ventilation during sleep. The weakening of the tone of the inspiratory and oropharyngeal muscles is one of the main causes of upper airways obstruction during the inspiratory phase.

DETAILED DESCRIPTION:
For patients with moderate OSAS, with few or no symptoms, without associated cardiovascular comorbidities, there is no recommended treatment. Rehabilitate the inspiratory and oropharyngeal muscles through muscle strengthening seems to be an alternative to this problem. Therefore, this study proposes a complete rehabilitation care evaluating the effectiveness of the strengthening of inspiratory and oropharyngeal muscles in subject with moderate OSAS.

ELIGIBILITY:
Inclusion Criteria:

* Moderate SAHOS (15 ≤ AHI ≤30);
* Body Mass Index (BMI) < 35 ;
* Patient affiliated or entitled to a social security scheme;
* Patient having signed a consent to participate in the study.

Exclusion Criteria:

* Excessive daytime sleepiness: Epworth sleepiness score > 10 ;
* Professional driving and history of accidents related to sleepiness;
* Severe obstructive or restrictive ventilatory disorders of neuromuscular origin authenticated by respiratory function tests;
* Patients undergoing treatment for OSAS or requiring immediate initiation of continuous positive airway pressure (CPAP) or a mandibular advancement orthosis;
* Patients who have stopped CPAP or orthosis treatment in less than one month;
* Patients undergoing cardiorespiratory exercise rehabilitation or starting regular physical training;
* Uncompensated heart failure, thoracic sternotomy surgery < 4 months;
* Marked osteoporosis with history of rib fractures;
* History of spontaneous pneumothorax;
* Severe asthma;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2024-12-30 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Apnea-Hypopnea Index (AHI) | At 3 months
  AHI is measured by polygraphy or polysomnography. It is not a score

SECONDARY OUTCOMES:
Maximum inspiratory pressure measurement (cmH2O) | At 3 and 9 Months
  Measured by POWERbreathe® K5
Neck circumference (cm) | At 3 months
  The neck circumference is measured by Magnetic Resonance Imagery (RMI)
Epworth sleepiness score | At 3 and 9 Months
  Sleep quality assessment using the Epworth sleepiness score. From 0 to 24. If score up to 10 then the patient has signs of excessive daytime sleepiness
Pittsburgh Sleep quality index | At 3 and 9 Months
  Sleep quality assessment using the Pittsburgh Sleep quality index. From 0 to 21. Score 0 = very good sleep quality. Score 21 = very poor sleep quality
Quality of life scale : Short Form 12 (SF12) | At 3 and 9 Months
  Quality of life assessment using the scale SF12 From 43 to 118 the higher the score, the better the quality of life
PICOT fatigue scale | At 3 and 9 Months
  Fatigue assessment using the PICOT scale From 0 to 32 If score up to 22 then the patient has signs of excessive sleepiness
AHI (Apnea-Hypopnea Index) | At 9 months
  AHI is measured by polygraphy or polysomnography It is not a score

CONTACTS AND LOCATIONS:
Overall Officials: Amandine Zellag, Principal Investigator — CHU SAINT-ETIENNE
Locations (2):
- France (2):
  - CHU de Grenoble, Grenoble
  - Centre Hospitalier Universitaire, Saint-Etienne